CLINICAL TRIAL: NCT04177940
Title: Denosumab (DMAB) Discontinuation and Switching in Glucocorticoid-Induced Osteoporosis (GIOP): a Pilot Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Maastricht University (Other); Vrije Universiteit Brussel (Other); Amgen (Industry)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300004179
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Denosumab (DMAB) to Alendronate (ALN) (Active Comparator): Switch from Denosumab 60 mg administered subcutaneously (SC) to weekly oral alendronate (70 mg; started 6 months after last denosumab dose)
  Interventions: Drug: DMAB Discontinuation and Switching
- DMAB to "Early" Zoledronic Acid (ZA) (Active Comparator): Switch from Denosumab 60 mg administered subcutaneously (SC) to one "early" zoledronic acid infusion (5 mg; 6 months after last denosumab dose)
  Interventions: Drug: DMAB Discontinuation and Switching
- DMAB to "Late" ZA (Active Comparator): Switch from Denosumab 60 mg administered subcutaneously (SC) to one "late" zoledronic acid infusion (5 mg; 9 months after last denosumab dose)
  Interventions: Drug: DMAB Discontinuation and Switching

INTERVENTIONS:
Drug: DMAB Discontinuation and Switching — Investigators will test the hypothesis that an increase in bone turnover markers (e.g. CTX and P1NP) in patients currently taking chronic glucocorticoids will be attenuated more in those who switch from denosumab to "late" zoledronic acid (9 months after last denosumab dose) compared to participants randomized to "early" zoledronic acid (6 months after last denosumab dose) or weekly alendronate (6 months after last denosumab dose

SUMMARY:
Investigators will test the hypothesis that an increase in bone turnover markers (e.g. carboxy-terminal collagen crosslinks (CTX) and P1NP) in patients currently taking chronic glucocorticoids will be attenuated more in those who switch from denosumab to "late" zoledronic acid (9 months after last denosumab dose) compared to participants randomized to "early" zoledronic acid (6 months after last denosumab dose) or weekly alendronate (6 months after last denosumab dose).

DETAILED DESCRIPTION:
This is an open-label, randomized, parallel-group pilot clinical trial in which Denosumab users will be assigned in a 1:1:1 allocation to one the following groups:

* Switch from Denosumab 60 mg administered subcutaneously (SC) to weekly oral alendronate (70 mg; started 6 months after last denosumab dose) OR
* Switch from Denosumab 60 mg administered subcutaneously (SC) to one "early" zoledronic acid infusion (5 mg; 6 months after last denosumab dose) OR
* Switch from Denosumab 60 mg administered subcutaneously (SC) to one "late" zoledronic acid infusion (5 mg; 9 months after last denosumab dose)

Participants will be advised to maintain adequate calcium and vitamin D intake per United States Department of Agriculture (USDA) and Department of Health and Human Services (DHHS) guidelines. All individuals will need ≥ 12 months of previous denosumab treatment (minimum of 2 doses) prior to switching to assigned randomization arm. The minimum number of doses (n = 2) is based on published data that the rebound in BMD might be less pronounced in patients receiving very limited denosumab. According to a systematic review of patients with multiple vertebral fractures following denosumab cessation, those with ≤2 years of denosumab treatment had fewer fractures compared with those with >2 years. Therefore, the maximum number of prior doses (n = 4) is based on higher incidence of rebound loss of bone mineral density (BMD), more rapid turnover, and potentially greater vertebral fractures after discontinuation of denosumab in patients who received more extensive treatment. Investigators will limit the trial to a more restricted use of denosumab duration (2-4 doses) to maintain greater homogeneity, given the somewhat smaller planned sample size. Users of denosumab will be sorted into two groups:

* Prevalent users: Defined as individuals with a minimum of one previous dose of denosumab, and up to 4 previous doses of denosumab (maximum). Prevalent users with one previous dose will receive a second dose of denosumab before proceeding to assigned randomization arm. Therefore, randomization will occur 2 weeks after screening visit if they had already 2-4 denosumab doses.
* New denosumab users: Defined as individuals who have not previously received denosumab. New users will receive two doses of denosumab before proceeding to assigned randomization arm.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, age 18 years or older and able to provide informed consent (IC)
* ≥ 3 months of glucocorticoid use at > 7.5 mg /day (prednisone equivalent dose) and anticipated to remain on glucocorticoids for at least six months
* A baseline BMD T-score of ≤ -2.0 at the lumbar spine, total hip, or femoral neck; OR
* A BMD T-score ≤ -1.0 at the lumbar spine, total hip, or femoral neck and a history of an osteoporotic fracture.

Exclusion Criteria:

* • Patients with fewer than three lumbar vertebrae that could be evaluated on dual energy x-ray absorptiometry (DXA)

  * Treatment with bisphosphonates in the preceding 2 years
  * Greater than 24 months (>4 injections) of prior treatment with denosumab
  * Women of childbearing potential, who are not currently using birth control, are pregnant, planning to become pregnant, or are breastfeeding. For women of childbearing potential: refusal to use 2 highly effective forms of contraception and to continue this practice for 7 months after last injection of study medication*
  * Men planning to conceive in the next 12 months
  * Unstable systemic medical condition
  * Uncontrolled hyperthyroidism
  * Uncontrolled hypothyroidism
  * History of Addison disease
  * History of osteomalacia
  * History of osteonecrosis of the jaw (ONJ)
  * History of atypical femur fracture
  * History of tooth extraction, jaw surgery, dental implants, or other dental surgery within the prior 6 months
  * History of anorexia nervosa, bulimia (by history or physical) or obvious malnutrition.
  * Invasive dental work(implants/surgery) planned in the next 2 years
  * History of Paget's disease of bone
  * Other bone diseases which affect bone metabolism
  * Vitamin D deficiency [25(OH) vitamin D level < 20 ng/mL (<49.9 nmol/L)]
  * Hypercalcemia >10% above upper limit of normal (ULN)
  * Elevated transaminases or total bilirubin ≥ 2.0 x ULN
  * History of any solid organ or bone marrow transplant
  * Malignancy within the last 5 years (except cervical carcinoma in situ or basal cell carcinoma or localized squamous cell carcinoma of the skin)
  * Hypocalcemia <10% below lower limit of normal (LLN)
  * Estimated glomerular filtration rate < 30 mL/minute/1.73 m^2
  * Intolerance to calcium supplements, vitamin D supplements
  * Contraindication to, or poorly tolerant of denosumab therapy (including hypersensitivity to the drug)
  * Contraindication to, or poorly tolerant of zoledronic therapy (including hypersensitivity to the drug)
  * Contraindication to, or poorly tolerant of alendronate (including hypersensitivity to the drug and sever gastro-intestinal intolerance to oral bisphosphonates)
  * Recipient of an investigational drug within 4 weeks prior to study drug administration
  * Not a good candidate for study participation in opinion of investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
CTX absolute difference V1 vs. V3 | 6 months post randomization
  Log of the absolute difference in CTX values between randomization (V1) and 6 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided